CLINICAL TRIAL: NCT07149831
Title: An Open-label, Single-center, Single-arm Phase I Clinical Trial Evaluating the Safety and Tolerability, Biodistribution and Radiation Dosimetry, and Pharmacokinetics of Flotufolastat F-18 Injection in Healthy Chinese Adults
Brief Title: A Clinical Trial Evaluating the Safety and Tolerability, Biodistribution and Radiation Dosimetry, and Pharmacokinetics of Flotufolastat F-18 Injection in Healthy Chinese Adults
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XTR020-101
Record Dates: First submitted 2025-08-04; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flotufolastat F-18 Injection (Experimental): Single dose 5.47~6.69mCi mCi intravenous injection of Flotufolastat F-18 Injection
  Interventions: Drug: Flotufolastat F-18 Injection

INTERVENTIONS:
Drug: Flotufolastat F-18 Injection — Single dose intravenous injection of Flotufolastat F-18 Injection . Serial whole-body PET scan will be obtain after injection, blood and urine collection after injection for the assessment of pharmacokinetics.

SUMMARY:
Flotufolastat F-18 Injection is a positron emission tomography (PET) imaging tracer that targets the extracellular domain of prostate-specific membrane antigen (PSMA). This phase I study investigated the safety, biodistribution, radiation dosimetry and Pharmacokinetics of Flotufolastat F-18 Injection in 6 healthy elderly Chinese volunteers.

DETAILED DESCRIPTION:
Flotufolastat F-18 Injection is a positron emission tomography (PET) imaging tracer that targets the extracellular domain of prostate-specific membrane antigen (PSMA). It is intended for the detection of prostate cancer (PCa) lesions.This Phase I study will be open-labeled, nonrandomized, single center study. Enrolled 6 healthy Chinese volunteers who meet all of the inclusion and none of the exclusion criteria. Subjects will receive 5.47~6.69mCi of Flotufolastat F-18 Injection via IV injection. Safety and tolerability will be observed. Biodistribution, pharmacokinetics, and dosimetry will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the content of study and voluntarily sign the informed consent form.
2. Healthy male or female, aged 18-60 (included).
3. Body mass index (BMI) between 19 and 26 kg/m² (included).
4. Vital signs, physical examination, 12-lead electrocardiogram (ECG), chest X-ray (posterior-anterior view), and abdominal ultrasound are normal, or any abnormalities that are diagnosed clinically insignificant.
5. Clinical laboratory test results are within normal ranges or any abnormalities that are diagnosed clinically insignificant.
6. Have the ability to communicate effectively with the investigator and comply with the study requirement to follow-up.
7. Female subject shouldcontracept effectively during the study period and 6 months after the study completed (effective contraception includes sterilization, intrauterine hormonal devices, condoms, contraceptive pills/agents, abstinence, or partner vasectomy). Male subject should agree to use contraception during the study period and 6 months after the study completed.

Exclusion Criteria:

1. Claustrophobia or inability to tolerate imaging examinations for any other reason.
2. Have a history of epilepsy or seizures, excluding childhood febrile seizures.
3. With chronic diseases, including but not limited to:

   1. cardiovascular, respiratory, gastrointestinal, urinary, hematological disease, neurological, endocrine, metabolic, or musculoskeletal diseases, or a history thereof.
   2. history of psychiatric disorders or currently significant psychiatric conditions
4. Have a history of asthma or allergies.
5. Have a history of malignant tumors.
6. Present any condition that may interfere with the absorption or metabolism of the investigational drug, or that may affect study results, as determined by the investigator to be clinically significant.
7. Underwent any surgical procedure within 3 months before administration or planned surgery during the study period.
8. Accomplished the blood donation or significant blood loss (>400 mL) within 3 months before administration or during the screening period.
9. Insufficient venous access (two distinct venous lines are required for investigational drug administration and PK sampling).
10. Known allergy to the active ingredient or any excipients of the investigational product.
11. Took any medications, including prescription, over-the-counter drugs, or herbal remedies, within 14 days before administration.
12. Participated any other new drug's clinical trial within 4 weeks prior to the administration or within 5 half-lives of the investigating drug (whichever is longer).
13. Radiopharmaceutical imaging or treatment within 7 days prior to screening or within 5 half-lives of the radiopharmaceutical (whichever is longer).
14. Pregnant or breastfeeding women.
15. Abnormal serological results (hepatitis B surface antigen, syphilis treponemal antibody, human immunodeficiency virus antibody, hepatitis C antibody) diagnosed clinically significant by the investigator.
16. QTc intervalis longer than 450 milliseconds during the screening period.
17. Major occupational exposure to ionizing radiation in the past 10 years (e.g., more than 50 mSv/year) or exposure to radioactive materials or ionizing radiation for therapeutic or research purposes.
18. Any reason determined by the investigator that could not complet the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Estimated)
Dates: Start 2025-06-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the biodistribution of Flotufolastat F-18 Injection after a single bolus intravenous injection in healthy Chinese adults. (%ID) | Day 1
  Radioactive accumulation (%ID) in target organs following administration of Flotufolastat F-18 Injection.
To evaluate the biodistribution of Flotufolastat F-18 Injection after a single bolus intravenous injection in healthy Chinese adults. | Day 1
  Standardized uptake value (SUV) in target organs following administration of Flotufolastat F-18 Injection.

SECONDARY OUTCOMES:
To assess the radiation dosimetry of Flotufolastat F-18 Injection | Day 1
  Radiation dose in target organs and whole-body effective dose following administration of Flotufolastat F-18 Injection
To evaluate the pharmacokinetic of Flotufolastat F-18 Injection | Day 1
  Radioactivity concentration (%ID/g) in whole blood, plasma, and urine samples at various time points post Flotufolastat F-18 Injection, and associated time activity curves.
Proportions of radioactive parent compound in plasma | Day 1
  To evaluate the pharmacokinetic of Flotufolastat F-18 Injection
To evaluate the safety profile of Flotufolastat F-18 Injection | Day 2
  Types, severity, incidence, and outcomes of adverse events (AEs) and serious adverse events (SAEs) reported during the study period

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No